CLINICAL TRIAL: NCT01624883
Title: The China PEACE (Patient-centered Evaluative Assessment of Cardiac Events Retrospective Study of Acute Myocardial Infarction
Brief Title: China PEACE-Retrospective AMI Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: WSGY-201202025-1
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary heart disease (CHD) and heart attacks pose a serious health risk to men and women, however the knowledge about the real-life AMI management in China is limited. Within a nation-wide and regional representative probability sample of hospitals in China, 27,800 AMI inpatient cases will be sampled randomly from 2001 to 2011. The sampled medical records will be reviewed and abstracted in the national coordinating centre, in order to evaluate the treatment pattern, outcomes, and cost for AMI patients, during the past decade. Basic data and innovative evidence will accelerate evidence-based clinical practice and policy making, and improve AMI patients outcomes finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. In addition, little information is available about the magnitude, prognosis, and optimal management of AMI, which is one of the leading causes of mortality and morbidity, both in rural and urban area. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

To investigate the treatment pattern and outcomes of AMI patients during the past decade in China, using a stratified two-stage cluster sampling design, from 175 sampled hospitals, 13,900 AMI cases will be selected in 2011, and 6,950 in 2001 and 2006 separately. Photocopies of the 27,800 medical records of AMI cases will be sent to the national coordinating centre. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted by well trained professional abstractors. By characterizing differences in patients' features, comparing the use of medications and procedures, and examining the in-hospital outcomes, we'll define the gaps between clinical practice and guidelines, as well as the disparities across different regions and hospitals, to evaluated the treatment pattern and outcomes in the last decade in China. New knowledge will be generated about AMI management all over China, to provide evidence for policy-making and clinical guidelines, and to improve AMI patients prognosis in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute myocardial infarction (AMI) according to discharge diagnosis (ICD-9 codes 410 or ICD-10 codes I21)

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using a stratified two-stage cluster sampling design, 175 hospitals will be selected from different regions in China, and 13,900 AMI inpatient cases will be selected in 2011, and 6,950 in 2001 and 2006 separately, from these sample hospitals.
Sampling Method: Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of all-cause death | Duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University

REFERENCES:
- [Derived] Guo W, Du X, Gao Y, Hu S, Lu Y, Dreyer RP, Li X, Spatz ES, Masoudi FA, Krumholz HM, Zheng X. Sex Differences in Characteristics, Treatments, and Outcomes Among Patients Hospitalized for Non-ST-Segment-Elevation Myocardial Infarction in China: 2006 to 2015. Circ Cardiovasc Qual Outcomes. 2022 Jun;15(6):e008535. doi: 10.1161/CIRCOUTCOMES.121.008535. Epub 2022 May 24. PMID 35607994
- [Derived] Wang X, Du X, Yang H, Bucholz E, Downing N, Spertus JA, Masoudi FA, Li J, Guan W, Gao Y, Hu S, Bai X, Krumholz HM, Li X. Use of intravenous magnesium sulfate among patients with acute myocardial infarction in China from 2001 to 2015: China PEACE-Retrospective AMI Study. BMJ Open. 2020 Mar 26;10(3):e033269. doi: 10.1136/bmjopen-2019-033269. PMID 32220910
- [Derived] Spatz ES, Wang Y, Beckman AL, Wu X, Lu Y, Du X, Li J, Xu X, Davidson PM, Masoudi FA, Spertus JA, Krumholz HM, Jiang L. Traditional Chinese Medicine for Acute Myocardial Infarction in Western Medicine Hospitals in China. Circ Cardiovasc Qual Outcomes. 2018 Mar;11(3):e004190. doi: 10.1161/CIRCOUTCOMES.117.004190. PMID 29848478
- [Derived] Qi Y, Wang W, Zhang K, An S, Wang S, Zheng J, Tang YD. Development and validation of Women Acute Myocardial Infarction in-Hospital Mortality Score (WAMI Score). Int J Cardiol. 2018 May 15;259:31-39. doi: 10.1016/j.ijcard.2017.12.010. PMID 29579607
- [Derived] Li X, Murugiah K, Li J, Masoudi FA, Chan PS, Hu S, Spertus JA, Wang Y, Downing NS, Krumholz HM, Jiang L; China PEACE Collaborative Group. Urban-Rural Comparisons in Hospital Admission, Treatments, and Outcomes for ST-Segment-Elevation Myocardial Infarction in China From 2001 to 2011: A Retrospective Analysis From the China PEACE Study (Patient-Centered Evaluative Assessment of Cardiac Events). Circ Cardiovasc Qual Outcomes. 2017 Nov;10(11):e003905. doi: 10.1161/CIRCOUTCOMES.117.003905. PMID 29158421
- [Derived] Murugiah K, Wang Y, Nuti SV, Li X, Li J, Zheng X, Downing NS, Desai NR, Masoudi FA, Spertus JA, Jiang L, Krumholz HM; China PEACE Collaborative Group. Are non-ST-segment elevation myocardial infarctions missing in China? Eur Heart J Qual Care Clin Outcomes. 2017 Oct 1;3(4):319-327. doi: 10.1093/ehjqcco/qcx025. PMID 28950309
- [Derived] Downing NS, Wang Y, Dharmarajan K, Nuti SV, Murugiah K, Du X, Zheng X, Li X, Li J, Masoudi FA, Spertus JA, Jiang L, Krumholz HM. Quality of Care in Chinese Hospitals: Processes and Outcomes After ST-segment Elevation Myocardial Infarction. J Am Heart Assoc. 2017 Jun 23;6(6):e005040. doi: 10.1161/JAHA.116.005040. PMID 28645937
- [Derived] Zhao S, Murugiah K, Li N, Li X, Xu ZH, Li J, Cheng C, Mao H, Downing NS, Krumholz HM, Jiang LX. Admission Glucose and In-hospital Mortality after Acute Myocardial Infarction in Patients with or without Diabetes: A Cross-sectional Study. Chin Med J (Engl). 2017 Apr 5;130(7):767-775. doi: 10.4103/0366-6999.202733. PMID 28345539
- [Derived] Li X, Li J, Masoudi FA, Spertus JA, Lin Z, Krumholz HM, Jiang L; China PEACE Collaborative Group. China PEACE risk estimation tool for in-hospital death from acute myocardial infarction: an early risk classification tree for decisions about fibrinolytic therapy. BMJ Open. 2016 Oct 24;6(10):e013355. doi: 10.1136/bmjopen-2016-013355. PMID 27798032
- [Derived] Li J, Li X, Hu S, Yu Y, Yan XF, Jiang LX. [ST-segment elevation myocardial infarction in the eastern urban China: from 2001 to 2011]. Zhonghua Xin Xue Guan Bing Za Zhi. 2016 Apr 24;44(4):303-8. doi: 10.3760/cma.j.issn.0253-3758.2016.04.006. Chinese. PMID 27112607
- [Derived] Du X, Spatz ES, Dreyer RP, Hu S, Wu C, Li X, Li J, Wang S, Masoudi FA, Spertus JA, Nasir K, Krumholz HM, Jiang L; China PEACE Collaborative Group. Sex Differences in Clinical Profiles and Quality of Care Among Patients With ST-Segment Elevation Myocardial Infarction From 2001 to 2011: Insights From the China Patient-Centered Evaluative Assessment of Cardiac Events (PEACE)-Retrospective Study. J Am Heart Assoc. 2016 Feb 22;5(2):e002157. doi: 10.1161/JAHA.115.002157. PMID 26903002
- [Derived] Zhang H, Masoudi FA, Li J, Wang Q, Li X, Spertus JA, Ross JS, Desai NR, Krumholz HM, Jiang L; China PEACE Collaborative Group. National assessment of early beta-blocker therapy in patients with acute myocardial infarction in China, 2001-2011: The China Patient-centered Evaluative Assessment of Cardiac Events (PEACE)-Retrospective AMI Study. Am Heart J. 2015 Sep;170(3):506-15.e1. doi: 10.1016/j.ahj.2015.05.012. Epub 2015 May 22. PMID 26385034
- [Derived] Zhang L, Desai NR, Li J, Hu S, Wang Q, Li X, Masoudi FA, Spertus JA, Nuti SV, Wang S, Krumholz HM, Jiang L; China PEACE Collaborative Group. National Quality Assessment of Early Clopidogrel Therapy in Chinese Patients With Acute Myocardial Infarction (AMI) in 2006 and 2011: Insights From the China Patient-Centered Evaluative Assessment of Cardiac Events (PEACE)-Retrospective AMI Study. J Am Heart Assoc. 2015 Jul 10;4(7):e001906. doi: 10.1161/JAHA.115.001906. PMID 26163041
- [Derived] Guan W, Murugiah K, Downing N, Li J, Wang Q, Ross JS, Desai NR, Masoudi FA, Spertus JA, Li X, Krumholz HM, Jiang L; China PEACE Collaborative Group. National quality assessment evaluating spironolactone use during hospitalization for acute myocardial infarction (AMI) in China: China Patient-centered Evaluation Assessment of Cardiac Events (PEACE)-Retrospective AMI Study, 2001, 2006, and 2011. J Am Heart Assoc. 2015 Jun 12;4(6):e001718. doi: 10.1161/JAHA.114.001718. PMID 26071031
- [Derived] Zhan L, Masoudi FA, Li X, Hu S, Venkatesh AK, Spertus JA, Lin Z, Desai NR, Li J, Krumholz HM, Jiang L; China PEACE Collaborative Group. Trends in cardiac biomarker testing in China for patients with acute myocardial infarction, 2001 to 2011: China PEACE-retrospective AMI study. PLoS One. 2015 Apr 20;10(3):e0122237. doi: 10.1371/journal.pone.0122237. eCollection 2015. PMID 25893247
- [Derived] Liu J, Masoudi FA, Spertus JA, Wang Q, Murugiah K, Spatz ES, Li J, Li X, Ross JS, Krumholz HM, Jiang L; China PEACE Collaborative Group. Patterns of use of angiotensin-converting enzyme inhibitors/angiotensin receptor blockers among patients with acute myocardial infarction in China from 2001 to 2011: China PEACE-Retrospective AMI Study. J Am Heart Assoc. 2015 Feb 23;4(2):e001343. doi: 10.1161/JAHA.114.001343. PMID 25713293
- [Derived] Zheng X, Dreyer RP, Hu S, Spatz ES, Masoudi FA, Spertus JA, Nasir K, Li X, Li J, Wang S, Krumholz HM, Jiang L; China PEACE Collaborative Group. Age-specific gender differences in early mortality following ST-segment elevation myocardial infarction in China. Heart. 2015 Mar;101(5):349-55. doi: 10.1136/heartjnl-2014-306456. Epub 2014 Dec 15. PMID 25510395
- [Derived] Gao Y, Masoudi FA, Hu S, Li J, Zhang H, Li X, Desai NR, Krumholz HM, Jiang L; China PEACE Collaborative Group. Trends in early aspirin use among patients with acute myocardial infarction in China, 2001-2011: the China PEACE-Retrospective AMI study. J Am Heart Assoc. 2014 Oct 10;3(5):e001250. doi: 10.1161/JAHA.114.001250. PMID 25304853
- [Derived] Li J, Li X, Wang Q, Hu S, Wang Y, Masoudi FA, Spertus JA, Krumholz HM, Jiang L; China PEACE Collaborative Group. ST-segment elevation myocardial infarction in China from 2001 to 2011 (the China PEACE-Retrospective Acute Myocardial Infarction Study): a retrospective analysis of hospital data. Lancet. 2015 Jan 31;385(9966):441-51. doi: 10.1016/S0140-6736(14)60921-1. Epub 2014 Jun 23. PMID 24969506
- [Derived] Dharmarajan K, Li J, Li X, Lin Z, Krumholz HM, Jiang L; China PEACE Collaborative Group. The China Patient-Centered Evaluative Assessment of Cardiac Events (China PEACE) retrospective study of acute myocardial infarction: study design. Circ Cardiovasc Qual Outcomes. 2013 Nov;6(6):732-40. doi: 10.1161/CIRCOUTCOMES.113.000441. Epub 2013 Nov 12. PMID 24221838